CLINICAL TRIAL: NCT03708445
Title: Development of a New Immunochemistry Method Using Antibodies of Aminoacyl-tRNA Synthetases Group and Aminoacyl-transfer Ribonucleic Acid Synthetases-interacting Multifunctional protein2 Lacking Exon 2 in the Bile Duct Cancer Cell; Multicenter Study
Brief Title: Development of a New Immunochemistry Method Using Antibodies of Proteins Related Bile Duct Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Collaborators: Korea Institute of Science and Technology (Other)
Responsible Party: Principal Investigator, Sung III Jang, Assistant professor, MD, PhD, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3-2016-0286
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Bile Duct Obstruction, Extrahepatic
Keywords: bile duct obstruction, extrahepatic; cytology; aminoacyl-tRNA synthetases
MeSH Terms: conditions — Cholestasis, Extrahepatic

STUDY DESIGN:
Intervention Model Description: The conventional staining method and new staining method will be performed in cytology specimens obtained from same patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bile duct stenosis (Experimental): This arm includes patients with bile duct stenosis. Endobiliary brushing cytology specimens will be obtained with endoscopic retrograde cholangiopancreatography (ERCP) of patients with bile duct stenosis. Cytology staining will be performed in the cytology specimens.
  Interventions: Diagnostic Test: Cytology staining

INTERVENTIONS:
Diagnostic Test: Cytology staining — Two staining will be performed in cytology specimens obtained from same patient. The cytology specimen will be obtained through brushing cytology using endoscopic retrograde cholangiopancreatography
  1. conventional cytology staining method
  2. new cytology staining method using antibody of aminoacyl-tRNA synthetases

SUMMARY:
The sensitivity of brushing cytology used to distinguish the cause of biliary strictures is low and clinical usefulness is not secured. The aim of this study was to develop a new differential staining method for cytology which is difficult to differentiate by the conventional staining method using biliary cancer related protein expressed only in bile duct cancer.

DETAILED DESCRIPTION:
Hypothesis: The statistical significance of new staining method using aminoacyl-tRNA synthetases (ARSs) group in normal bile duct cells and the bile duct cancer cells collected by endoscopic retrograde pancreaticoduodenoscopy (ERCP) will be compared to prove the usefulness of the new staining method.

Clinical study design: The bile duct cytology will be obtained by brushing cytology using ERCP in patients with biliary stenosis. The expression of ARSs in the brushing cytology will be evaluated by new staining method and compare with the results of conventional cytology staining method including Papanicolaou staining. Immunofluorescence or immunohistochemistry staining will be performed to differentiate the presence of the tumor. The sensitivity and specificity of the new staining method will be compared with the conventional staining method and its usefulness be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biliary cancer confirmed by imaging (CT, MRI, positron emission tomography)
* Patients with bile duct cancer diagnosed using brushing cytology by endoscopic retrograde pancreaticoduodenoscopy
* Patients who underwent surgical treatment with biliary cancer
* Patients with bile duct stenosis

Exclusion Criteria:

* Minors under the age of 19, vulnerable subjects such as illiteracy
* Necrotic specimens
* Samples with non-diagnostic cytology results and insufficient cells for further evaluation
* Samples classified as neoplastic (benign or other)
* Patient with cholangitis in the bile duct

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
The usefulness of new staining method | 1 year
  The sensitivity, specificity, positive predictive value, negative predictive value and accuracy of new staining method will be compared with th conventional Pap staining of brushing cytology specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Institutional Review Board, Study Chair — Gangnam Severance Hospital, Yonsei University College of Medicine
Locations (6):
- South Korea (6):
  - CHA Bundang Medical Center, Seongnam, Bundang-gu
  - Gangnam Severance Hospital, Seoul, Gangnam-gu
  - In Ha University Hospital, Incheon, Jung-gu
  - Soon Chun Hyang University Hospital, Cheonan, Cheonan, Namdong-gu
  - Gachon University Gil Medical Center, Incheon, Namdong-gu
  - Pusan National University Hospital, Busan, Seo-gu

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the following individual participant data with other researchers during study period.
  Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR), Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: * Primary investigator
  * Sub primary investigator

REFERENCES:
- [Derived] Jang SI, Nahm JH, Kwon NH, Jeong S, Lee TH, Cho JH, Kwon CI, Kim DU, Kim JM, Cho HD, Lee HS, Kim S, Lee DK. Clinical utility of methionyl-tRNA synthetase 1 immunostaining in cytologic brushings of indeterminate biliary strictures: a multicenter prospective study. Gastrointest Endosc. 2021 Oct;94(4):733-741.e4. doi: 10.1016/j.gie.2021.04.026. Epub 2021 May 6. PMID 33965384